CLINICAL TRIAL: NCT04890652
Title: Digital Interventions to Treat Hazardous Drinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000026333; R01AA026844-02S1 (NIH)
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Hazardous Drinking; Stress
Keywords: Hazardous drinking; COVID-19; Stress; Digital intervention
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: All participants received a 4-week digital intervention, "Emotion regulation via Breathing for Alcohol reduction (EBA)," which combines alcohol intervention with stress reduction techniques based on self-regulated breathing exercises. The preliminary efficacy of this digital intervention was evaluated through assessments conducted before and immediately after the intervention, as well as during a follow-up assessment 30 days later.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Risky drinkers (Other): All participants will receive the same 4-week intervention program.
  Interventions: Behavioral: Digital intervention

INTERVENTIONS:
Behavioral: Digital intervention — All participants will receive a digital intervention designed to reduce stress and alcohol consumption over a 4-week period. The intervention will include two weekly sessions that integrate alcohol intervention with breathing-based stress management techniques.

SUMMARY:
There has been a significant increase in the prevalence of stress- and alcohol- related disorders during the COVID-19 pandemic. This project aims to conduct a feasibility study to evaluate the preliminary efficacy of a digital intervention designed to reduce stress and alcohol use. Additionally, this study will examine the impact of stress, including COVID-19 related stress, on the risk of alcohol misuse and the outcomes of the intervention in risky social drinkers.

DETAILED DESCRIPTION:
This project proposes a feasibility study to evaluate the preliminary efficacy of a digital intervention aimed at addressing stress-related drinking in risky drinkers with emotional stress. This digital intervention combines telehealth- and smartphone app- based approaches, allowing concurrent intervention and participant-initiated daily exercise in a real-life setting. This program integrates alcohol intervention with breathing-based stress reduction and focuses on developing emotion regulation skills to manage stress, craving, and alcohol misuse. After the 4-week intervention, all participants will be prospectively followed for 30 days to monitor stress, alcohol use, and other health-related behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Heavy or binge drinkers
* Either high or low COVID-19 related stress

Exclusion Criteria:

* Current or past substance use disorder other than mild alcohol, tobacco, marijuana use disorder
* Psychiatric disorders except for mood and anxiety disorders
* Any significant current medical conditions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dongju Seo, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited starting on October 13, 2021 via online platforms (e.g., craigslist) and flyers. A recruitment center was located in New Haven, Connecticut.
Pre-assignment Details: Out of the 33 enrolled participants, six participants did not start the study due to scheduling difficulties (N=2), no shows (N=3), and obtaining a new job (N=1).
Groups:
- Digital Intervention (4-week): All participants received a 4-week digital intervention, "Emotion regulation via Breathing for Alcohol Reduction (EBA)," which combines alcohol intervention with stress reduction techniques based on self-regulated breathing exercises. The preliminary efficacy of this digital intervention was evaluated through assessments conducted before and immediately after the intervention, as well as during a follow-up assessment 30 days later.
Period: Overall Study
Arm/Group | Digital Intervention (4-week)
Started | 27
Completed | 25
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Digital Intervention (4-week): All participants received a 4-week digital intervention, "Emotion regulation via Breathing for Alcohol Reduction (EBA)," which combines alcohol intervention with stress reduction techniques based on self-regulated breathing exercises. The preliminary effects of this digital intervention were evaluated through assessments conducted before and immediately after the intervention, as well as during a follow-up assessment 30 days later.
Arm/Group | Digital Intervention (4-week)
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in Alcohol Use (Quantity)
Description: The average number of alcoholic beverages consumed per week (drinks per week), as measured by the Timeline Follow Back.
Time Frame: baseline, immediately post-intervention, and follow-up (30 days)
Population: Two participants (N=2) discontinued participation in the study following the baseline assessment; One participant withdrew during the second week of the intervention due to scheduling difficulties from a personal busy schedule, and the other participant withdrew in week 4 of the intervention due to non-compliance issues (e.g., repeated instances of not showing up).
Measure: Mean (Standard Deviation); unit: drinks per week
Groups:
- Digital Intervention: Participants received a 4-week digital intervention, "Emotion regulation via Breathing for Alcohol Reduction (EBA)." Alcohol use outcomes were evaluated through assessments conducted before and immediately after the intervention, as well as during a follow-up assessment 30 days later.
Arm/Group | Digital Intervention
Number analyzed (Participants) | 27
drinks per week
  Baseline | 15.4 (13.0)
  Immediately Post-intervention: number analyzed (Participants) | 25
  Immediately Post-intervention | 8.5 (8.1)
  30 day follow up: number analyzed (Participants) | 25
  30 day follow up | 7.5 (7.8)
Statistical Analysis 1: Comparison: Digital Intervention; Test type: Other — single group. The power-related information was estimated by calculating the effect size, specifically partial eta squared; p < 0.001, General Linear Model

2. Primary Outcome: Change in Alcohol Use (Frequency)
Description: The number of drinking days per week, as measured by the Timeline Follow Back.
Time Frame: baseline, immediately post-intervention, follow-up (30 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: drinking days per week
Arm/Group | Digital Intervention
Number analyzed (Participants) | 27
drinking days per week
  baseline | 4.5 (2.2)
  immediately post-intervention: number analyzed (Participants) | 25
  immediately post-intervention | 2.9 (1.9)
  30 day follow-up: number analyzed (Participants) | 25
  30 day follow-up | 2.7 (2.3)
Statistical Analysis 1: Comparison: Digital Intervention; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, General Linear Model

ADVERSE EVENTS:
Time Frame: 2.5 months
Groups:
- Digital Intervention: All participants received a 4-week digital intervention, "Emotion regulation via Breathing for Alcohol Reduction (EBA)," which combines alcohol intervention with stress reduction techniques based on self-regulated breathing exercises. The preliminary efficacy of this digital intervention was evaluated through assessments conducted before and immediately after the intervention, as well as during a follow-up assessment 30 days later.
Arm/Group | Digital Intervention
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 3/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digital Intervention (N=27)
General disorders and administration site conditions - Other, specify (Infections and infestations) | 1 (1) — One episode of a respiratory infection, unrelated to the intervention, during the second week of the intervention.
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — One episode of cold symptoms, unrelated to the intervention, occurred during the first week of the intervention.
General disorders and administration site conditions - Other, specify (Nervous system disorders) | 1 (1) — One episode of moderate seizure-like symptoms, inherent to the participant and unrelated to the intervention, occurred post-intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT04890652/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT04890652/ICF_001.pdf